CLINICAL TRIAL: NCT03352895
Title: The Effects of Resveratrol on the Complications of Patients With Hemodialysis: a Prospective, Randomized, Double-blinded Clinical Trial
Brief Title: The Effects of Resveratrol on the Complications of Patients With Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dalin Tzu Chi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: B10401008
Record Dates: First submitted 2017-02-07; First posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-10

CONDITIONS: Chronic Kidney Disease
Keywords: Resveratrol; chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Resveratrol; Grape Seed Extract; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- control (Placebo Comparator): Control group will receive placebo medication therapy
  Interventions: Dietary Supplement: Placebo
- test group (Experimental): resveratrol group will receive oral resveratrol (100 mg per day)
  Interventions: Dietary Supplement: resveratrol

INTERVENTIONS:
Dietary Supplement: resveratrol — Grape seed extract 100mg Microcrystalline Cellulose 90mg Magnesium Stearate 2mg Gelatin 100mg
  Other Names: Grape seed extract
  Arms: test group
Dietary Supplement: Placebo — The gel contains a mixture of glucose and maltodextrin - a complex carbohydrate - along with fat and a trace of protein.
  Other Names: Maltodextrin
  Arms: control

SUMMARY:
Participants'll include 140 adult patients with CKD and receiving hemodialysis in our hospital, and divided them into 2 groups. Control group will receive placebo medication therapy; resveratrol group will receive oral resveratrol (100 mg per day). All participants will receive either treatment for 1year, and receive examinations of pure tone audiometry, speech reception thresholds, and speech discrimination score.

DETAILED DESCRIPTION:
Patients with chronic kidney disease (CKD) often suffered from hearing impairment, vertigo/dizziness, cognitive degeneration, cardiovascular diseases. In addition, compared to patients without CKD, the longevity of patients with CKD was also shorter. The mechanism underlying the complications of CKD were very complicated, but were generally associated with uremic toxins, tissue hypoxia, free radicals damages. Meanwhile, some co-morbidities, for example, diabetes mellitus, hypertension, atherosclerosis, would also worsen the complications of CKD. However, only limited methods were reported to have beneficial effects on renal function and its complications. For, example, controlling co-morbidities of CKD, avoiding nephrotoxic substances, and dialysis.

Resveratrol, it could prevent deterioration of cardiovascular diseases and cancer progression. But, the beneficial effects of resveratrol on hearing impairment, tinnitus, vertigo/dizziness, cognitive degeneration, cancer development, death in patients with CKD were also unclear.

This study aimed to investigate the beneficial effects of resveratrol on hearing impairment in patients with CKD by a prospective, randomized, double-blinded clinical trial design.

Participants'll include 140 adult patients with CKD and receiving hemodialysis in our hospital, and divided them into 2 groups. Control group will receive placebo medication therapy; resveratrol group will receive oral resveratrol (100 mg per day). All patients will receive either treatment for 1year, and receive examinations of pure tone audiometry, speech reception thresholds, and speech discrimination score.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic kidney disease (CKD) and routine hemodialysis
* Age limits 40~69 years old
* Normal hearing or symmetrical sensorineural hearing loss, all ears frequency differences are less than 15 dB

Exclusion Criteria:

* Life can not take care of themselves or the bed of a patient
* Acceptance of peritoneal dialysis patients
* Moderate hearing loss (pure tone average hearing threshold greater than 50 dB)
* Moderate or severe cognitive impairment (Mini-Mental State Examination score less than 21 points)
* The details of the study can not understand or can not fit the patient examination.
* A history of alcohol or drug abuse
* The high ambient noise exposure history
* Poor guide backbone pure tone hearing thresholds greater than 10 decibels, trying to listen to 4 kilohertz air conduction threshold is greater than 8 kilohertz air conduction threshold value of 20 dB
* Before the age of 30 have hearing loss
* Had a stroke, myocardial infarction, a history of cancer
* Pregnant woman

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Pure tone audiometry (PTA) | one year
  pure tone thresholds of 250, 500, 1000, 2000, 4000, 8000 Hz were measured.

SECONDARY OUTCOMES:
Speech Audiometry | one year
  Speech reception thresholds and speech discrimination scores were tested.

CONTACTS AND LOCATIONS:
Overall Officials: Juen-Haur Hwang, MD, PhD., Study Chair — Dalin Tzu Chi Hospital
Locations (1):
- Dalin Tzu Chi Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided